CLINICAL TRIAL: NCT01262001
Title: A Phase 2, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Efficacy of FG-3019 in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: Safety, Tolerability, and Efficacy Study of Idiopathic Pulmonary Fibrosis
Acronym: FGCL-3019-049
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-3019-049
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pamrevlumab

STUDY DESIGN:
Intervention Model Description: FG-3019 administered at dose of 15 mg/kg (Cohort 1 ) by IV infusion every 3 weeks for 45 weeks in the target population.(first treatment year and first extended treatment year) and every 3 weeks thereafter for three additional extended treatment years.
Masking Description: FG-3019 administered at dose of 30 mg/kg (Cohort 2 ) by IV infusion every 3 weeks for 45 weeks in the target population.(first treatment year and first extended treatment year) and every 3 weeks thereafter for three additional extended treatment years.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1/1-EX (Experimental): Subjects with moderate to severe idiopathic pulmonary fibrosis (IPF) who have evidence of disease progression
  Interventions: Drug: FG-3019
- Cohort 2/2-EX (Experimental): Subjects with mild to moderate idiopathic pulmonary fibrosis (IPF) who have evidence of disease progression
  Interventions: Drug: FG-3019

INTERVENTIONS:
Drug: FG-3019 — Cohort 1 and Cohort 1-EX: 15 mg/kg by infusion every 3 weeks for 45 weeks in the target population (first treatment year and first extended treatment year and every 3 weeks thereafter for three additional extended treatment years).
  Other Names: Pamrevlumab
  Arms: Cohort 1/1-EX
Drug: FG-3019 — Cohort 2 and Cohort 2-EX: 30 mg/kg by infusion every 3 weeks for 45 weeks in the target population (first treatment year and first extended treatment year and every 3 weeks thereafter for three additional extended treatment years).
  Other Names: Pamrevlumab
  Arms: Cohort 2/2-EX

SUMMARY:
To evaluate the safety and tolerability of FG-3019 in subjects with Idiopathic Pulmonary Fibrosis (IPF) and the efficacy of FG-3019 for attenuating fibrosis in these subjects.

DETAILED DESCRIPTION:
Major Changes: FGCL-3019-049 Protocol Amendment 3 offers long-term extension of treatment with FG-3019 to eligible Cohort 1-EX (approximately 14 subjects) and Cohort 2 (approximately 28 subjects) subjects who complete the Week 48-EX and Week 48 assessments described in Protocol Amendment 2, respectively. A subject is eligible for long-term extension of treatment if the investigator, after discussion with the Fibrogen Medical Monitor, believes that the subject would benefit from continued treatment with FG-3019.

ELIGIBILITY:
Main Inclusion Criteria:

1. Age 35 to 80 years, inclusive.
2. Clinical diagnosis of IPF by high resolution computed tomography (HRCT) scan (and in some cases by surgical lung biopsy) and reduced lung function (forced vital capacity).
3. History of IPF of 5 years duration or less.
4. Evidence of progression of IPF within the last 3-12 months for Cohort 1, or within the last 18 months for Cohort 2 before screening.
5. Women of childbearing potential, and men, must be willing to use a medically acceptable method of contraception during the trial and 3 months after the last dose of study drug.

Main Exclusion Criteria:

1. Women who are pregnant or nursing.
2. History of any other types of lung or heart disease and any other medical conditions that, in the opinion of the investigator, would preclude the subject's participation in the study.
3. Clinically important abnormal laboratory tests.
4. Upper or lower respiratory tract infection of any type within 4 weeks of the first screening visit.
5. Acute exacerbation of IPF within 3 months of the first screening visit.
6. Use of certain medications within 4 weeks of the first screening visit.
7. Receipt of an investigational drug within 6 weeks of the first screening visit.
8. History of cancer of any type in the 5 years preceding the first screening visit, excluding non-melanomatous skin cancer, localized bladder cancer, or in situ cervical cancer.
9. Trauma or surgical procedures requiring hospitalization within 4 weeks of the first screening visit.
10. Planned elective surgery during the study including 4 weeks following the final dose of study drug.
11. History of allergic or anaphylactic reaction to human, humanized, chimeric or murine monoclonal antibodies.
12. Inability to cooperate with study personnel or history of non-compliance to a medical regimen.
13. Previous treatment with FG-3019.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-03; Primary Completion 2014-06-26 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of FG-3019 administered at doses of 15 mg/kg (Cohort 1 and Cohort 1-EX) and 30 mg/kg (Cohort 2 and Cohort 2-EX) every 3 wks for 45 weeks, and every 3 weeks thereafter for three additional treatment years. | Cohort 1: Up to 60 weeks, Cohort 1-EX (original subjects): up to 109 weeks, Cohort 1-EX (subjects who complete Week 48-EX and continue in the trial): up to 151 weeks, Cohort 2: up to 58 weeks, Cohort 2-EX: up to 202 weeks

SECONDARY OUTCOMES:
To evaluate the effect of FG-3019 on the extent of pulmonary fibrosis in subjects with IPF. | Cohort 1: Up to 60 weeks, Cohort 1-EX (original subjects): up to 109 weeks, Cohort 1-EX (subjects who complete Week 48-EX and continue in the trial): up to 151 weeks, Cohort 2: up to 58 weeks, Cohort 2-EX: up to 202 weeks
To evaluate the effect of FG-3019 on pulmonary function in subjects with IPF. | Cohort 1: Up to 60 weeks, Cohort 1-EX (original subjects): up to 109 weeks, Cohort 1-EX (subjects who complete Week 48-EX and continue in the trial): up to 151 weeks, Cohort 2: up to 58 weeks, Cohort 2-EX: up to 202 weeks
To evaluate the effect of FG-3019 on dyspnea in subjects with IPF. | Cohort 1: Up to 60 weeks, Cohort 1-EX (original subjects): up to 109 weeks, Cohort 1-EX (subjects who complete Week 48-EX and continue in the trial): up to 151 weeks, Cohort 2: up to 58 weeks, Cohort 2-EX: up to 202 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Arizona Pulmonary Specialists, LTD, Scottsdale, Arizona
  - Yale University, New Haven, Connecticut
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Via Christi Hospitals Wichita, Inc., Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - St. Luke's Hospital, Chesterfield, Missouri
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Mount Sinai, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah - Lung Health Research, Salt Lake City, Utah
  - Vermont Lung Center, Colchester, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - University of Wisconsin School of Medicine & Public Health, Madison, Wisconsin

REFERENCES:
- [Derived] Kim GH, Zhang X, Brown MS, Poole L, Goldin J. Minimum clinically important difference in Quantitative Lung Fibrosis score associated with all-cause mortality in idiopathic pulmonary fibrosis: subanalysis from two phase II trials of pamrevlumab. BMJ Open. 2025 May 12;15(5):e094559. doi: 10.1136/bmjopen-2024-094559. PMID 40355288
- [Derived] Raghu G, Scholand MB, de Andrade J, Lancaster L, Mageto Y, Goldin J, Brown KK, Flaherty KR, Wencel M, Wanger J, Neff T, Valone F, Stauffer J, Porter S. FG-3019 anti-connective tissue growth factor monoclonal antibody: results of an open-label clinical trial in idiopathic pulmonary fibrosis. Eur Respir J. 2016 May;47(5):1481-91. doi: 10.1183/13993003.01030-2015. Epub 2016 Mar 10. PMID 26965296